CLINICAL TRIAL: NCT07260240
Title: Comparison of the Efficacy of Intravenous Fluid Administration Between Bolus and Continuous Infusion in Pregnant Women With Fetal Heart Rate Tracing Category II: A Randomized Controlled Trial
Acronym: Bolus fluid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 013/2568
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Fetal Non Reassuring
Keywords: Bolus fluid administration, Non-reassuring fetal status, Fetal distress, Intrauterine resuscitation
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups using computer-generated block 0f-four randomization. The experimental group receives 500 mL of normal saline intravenously as a bolus in 30 minutes, followed by 1,000 mL normal saline at 150 mL/hour, while the control group receives 1,000 mL of normal saline at 150 mL/hour without a preceding bolus.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Bolus group): Receives 500 mL of normal saline intravenously as a bolus (Experimental): Receives 500 mL of normal saline intravenously as a bolus over 20 minutes, followed by 1,000 mL normal saline at 150 mL/hour
  Interventions: Drug: Giving 500 mL of normal saline intravenously as a bolus over 20 minutes, followed by 1,000 mL normal saline at 150 mL/hour
- Group B (Continuous infusion group): Receives 1,000 mL of normal saline at 150 mL/hour (Experimental): Group B (Continuous infusion group): Receives 1,000 mL of normal saline at 150 mL/hour without a preceding bolus
  Interventions: Drug: Giving 500 mL of normal saline intravenously as a bolus over 20 minutes, followed by 1,000 mL normal saline at 150 mL/hour

INTERVENTIONS:
Drug: Giving 500 mL of normal saline intravenously as a bolus over 20 minutes, followed by 1,000 mL normal saline at 150 mL/hour — Giving 500 mL of normal saline intravenously as a bolus over 20 minutes, followed by 1,000 mL normal saline at 150 mL/hour which the another one will be giving 1,000 mL of normal saline at 150 mL/hour without a preceding bolus.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two methods of intravenous (IV) fluid administration-bolus infusion versus continuous infusion-for intrauterine resuscitation in pregnant women who present with Category II fetal heart rate (FHR) tracings during labor. The main research question is:

Does intrauterine resuscitation using an adjusted IV hydration bolus of normal saline more effectively convert the FHR tracing from Category II to Category I within 30 minutes compared to adjusted IV hydration using a continuous infusion of 1000 mL normal saline at 150 mL/hour? Objectives

Primary Objective:

- To compare the rate of improvement of electronic fetal monitoring (EFM) category from Category II to Category I within 30 minutes between two hydration methods: Normal saline bolus loading (adjusted dose) Normal saline continuous infusion (1000 mL at 150 mL/hr)

Secondary Objectives:

* To identify the characteristics of IV fluid administration used during intrauterine resuscitation.
* To determine whether fluid bolus improves fetal heart rate patterns more rapidly or effectively than continuous infusion.

Methods

Study Design: Randomized controlled trial with block randomization (block of four).

Participants: Pregnant women in labor who present with Category II FHR tracing on admission.

Intervention:

Group A: Adjusted IV hydration with normal saline bolus loading. Group B: Adjusted IV hydration with normal saline continuous infusion (1000 mL at 150 mL/hr).

Monitoring: Electronic fetal monitoring (EFM) will be continuously observed to detect any change in FHR category after intervention.

Primary Outcome: Conversion of FHR from Category II to Category I within 30 minutes.

DETAILED DESCRIPTION:
This is a randomized controlled trial study to compare the efficacy of two methods of intravenous (IV) fluid administration-bolus infusion versus continuous infusion-for intrauterine resuscitation in pregnant women who present with Category II fetal heart rate (FHR) tracings during labor

There are 2 interventions :

Intervention 1 (Bolus Group):

Participants receive 500 mL of normal saline (NSS) intravenously as a bolus over 20 minutes, followed by 1,000 mL of NSS infused continuously at 150 mL/hour.

Intervention 2 (Continuous Infusion Group):

Participants receive 1,000 mL of normal saline infused continuously at 150 mL/hour without a preceding bolus.

Short-term Outcome Collection

Primary short-term outcome:

Conversion of FHR Category II to Category I within 30 minutes after starting the assigned IV hydration regimen, assessed by continuous electronic fetal monitoring (EFM).

Secondary short-term outcomes:

Measured at baseline, 10 minutes, and 30 minutes after intervention:

Maternal hemodynamic parameters: Blood pressure, heart rate, respiratory rate, SpO₂ IVC collapsibility index (IVC-CI) assessed by ultrasound (M-mode) Umbilical artery Doppler indices: Resistance Index (RI), Pulsatility Index (PI), S/D ratio FHR variability and deceleration pattern All outcomes are recorded in the Case Record Form (CRF) by blinded assessors. All participants are women in labor with Category II fetal heart rate (FHR) tracing, randomized by block randomization (block size = 4).

During the intervention, standard intrauterine resuscitation measures (maternal left lateral position, discontinuation of oxytocin, oxygen 15 L/min by mask if indicated) are maintained uniformly.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton
2. Thai nationality
3. Gestational Age more than equal 37 Weeks
4. Maternal Age 20-35 Years
5. Cephalic Presentation
6. Electronic Fetal Monitoring (EFM) Category II

Exclusion Criteria:

1. Maternal underlying diseases : Cardiac disease, Pulmonary disease), Overt DM, Thyroid disease,. etc
2. High risk pregnancy :Pre-eclampsia/Eclampsia), GDM
3. Fetal abnormalities
4. Maternal receiving medications for example : Magnesium sulfate, Pethidine, Opioids
5. Oligohydramnios

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of improvement of electronic fetal monitoring (EFM) category from Category II to Category I within 30 minutes | 30 minutes
  To compare the rate of improvement of electronic fetal monitoring (EFM) category from Category II to Category I within 30 minutes between two hydration methods:
  1. Normal saline bolus loading (adjusted dose)
  2. Normal saline continuous infusion (1000 mL at 150 mL/hr)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Chon Buri 20110 Recruiting, Si Racha, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was saved in form of Microsoft excel spreadsheet and SPSS file